CLINICAL TRIAL: NCT00003433
Title: A Phase I/II Study of Active Immunotherapy With Carcinoembryonic Antigen RNA-Pulsed, Autologous, Cultured Dendritic Cells After Complete Resection of Hepatic Metastases of Colorectal Carcinoma
Brief Title: Immunotherapy in Treating Patients With Resected Liver Metastases From Colon Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066459; DUMC-2031-00-11R3; DUMC-2176-99-12R2; DUMC-97146; NCI-G98-1456
Record Dates: First submitted 1999-11-01; First posted 2003-08-13 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2002-11

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms

INTERVENTIONS:
Biological: carcinoembryonic antigen RNA-pulsed DC cancer vaccine

SUMMARY:
RATIONALE: Immunotherapy using CEA-treated white blood cells may help a person's body build an immune response to kill their tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of immunotherapy with CEA-treated white blood cells in treating patients with resected liver metastases from colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the cellular immune response to carcinoembryonic antigen pulsed dendritic cells in patients with adenocarcinoma of the colon metastatic to the liver.
* Evaluate the overall and recurrence free survival in this patient population.

OUTLINE: Patients undergo leukapheresis for up to 4.5 hours to collect dendritic cells. The separated dendritic cells are pulsed with carcinoembryonic antigen (CEA) RNA. Patients receive CEA RNA pulsed dendritic cells intravenously every 2 weeks for a total of 4 doses. Patients undergo a second leukapheresis 2 weeks after the last dendritic cell infusion to obtain specimens for immunologic tests. Patients with extra doses of dendritic cells available may receive additional doses of CEA RNA pulsed dendritic cells every 2 months in the absence of unacceptable toxicity.

Patients are followed at weeks 12, 24, 36, and 48, and every 6 months thereafter.

PROJECTED ACCRUAL: A total of 22 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon metastatic to the liver that expresses carcinoembryonic antigen (CEA) after resection with curative intent

  * At least 50% of the tumor cells must stain positive for CEA with at least moderate intensity
* No gross residual disease after surgery

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Greater than 6 months

Hematopoietic:

* Absolute neutrophil count at least 1000/mm 3
* Hemoglobin at least 9 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* No chronic or acute hepatic disease

Renal:

* Creatinine less than 2.5 mg/dL

Cardiovascular:

* No chronic or acute cardiac disease (New York Heart Association class III or IV)

Pulmonary:

* No chronic or acute pulmonary illness such as asthma or chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* No other prior or concurrent malignancy except nonmelanoma skin cancer or controlled superficial bladder cancer within the past 5 years
* No history of autoimmune disease such as inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, and multiple sclerosis
* No active acute or chronic infection such as urinary tract infection, HIV, or viral hepatitis
* No active infectious enteritis or eosinophilic enteritis

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No other concurrent immunotherapy

Chemotherapy:

* No concurrent chemotherapy
* At least 6 weeks since prior chemotherapy

Endocrine therapy:

* No concurrent steroid therapy (or any other immunosuppressives)
* At least 6 weeks since prior steroid therapy

Radiotherapy:

* No concurrent radiotherapy
* At least 6 weeks since prior radiotherapy

Surgery:

* Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert K. Lyerly, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States